CLINICAL TRIAL: NCT05519774
Title: Assessment of Cancer Related Brain Fog Using the Test of Strategic Learning
Acronym: ACT I
Status: Completed | Type: Observational
Sponsor: Inova Health Care Services (Other)
Collaborators: The University of Texas at Dallas (Other)
Responsible Party: Sponsor
Other Study IDs: U21-08-4519
Record Dates: First submitted 2022-08-11; First posted 2022-08-29 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Brain Fog
Keywords: Breast cancer
MeSH Terms: conditions — Mental Fatigue; Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Inova research team will ask people who have had an experience of breast cancer and related changes to their cognition to complete some scales that researchers have established describe brain fog (called patient reported outcomes) and compare those results to the TOSL results. This will be done twice to see if changes are detected similarly on both types of measures.

DETAILED DESCRIPTION:
Current brain fog research struggles to clearly define and measure brain fog because the changes are more subtle than typically show up on "objective" tests. These subtle changes on the tests, may not appear subtle in everyday life. This disconnect can lead to people managing cancer feeling unheard or unbelieved about their experience with brain fog. However, cognitive research outside of the cancer population has developed and tested tests that are more sensitive to cognitive changes and improvements. The goal of this initial research project is to test a more sensitive test, called the Test of Strategic Learning (TOSL), to see if it is sensitive enough to objectively measure brain fog.

One other problem with previous brain fog research is that it has not included a diverse population. Therefore, what we think we know about brain fog may not be true for everyone with brain fog. The diverse population in the DMV area that Inova serves deserves to have their experiences represented in the research.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* ECOG performance status ≤ 2
* Patients diagnosed or with a history of breast cancer within the last 5 years.
* Life expectancy of at least 3 months
* Subject reports experiencing brain fog or cognitive impairment that the subject attributes to cancer or cancer therapy
* Able to sit for one hour and attend and respond to verbal and written instructions.
* Able to use a computer

Exclusion Criteria:

* Brain metastases from breast cancer
* Severe hearing or visual impairment
* Unable to give informed consent
* Unable to read and write in English
* Those diagnosed with history of neurologic injuries or disorders (e.g. seizures, strokes, traumatic brain injury, brain surgery, neurodegenerative disorders) other than those attributable to cancer or cancer therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men or women with stage I-III breast cancer.
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-10-18 (Actual)

PRIMARY OUTCOMES:
Number of months to recruit | 4 months
  Number of months between opening of recruitment and recruitment date of the 10th subject.
Correlation between the TOSL score and PAOFI score | 6 months
  Spearman correlation coefficient between the TOSL Lessons score and the PAOFI higher level cognition subscale score.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Cohen, MD, Principal Investigator — Inova Health Care Services
Locations (1):
- Inova HCS, Falls Church, Virginia, United States

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-20): https://cdn.clinicaltrials.gov/large-docs/74/NCT05519774/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-28): https://cdn.clinicaltrials.gov/large-docs/74/NCT05519774/ICF_001.pdf